CLINICAL TRIAL: NCT00516113
Title: A Placebo-Controlled Study to Investigate the Onset of Action of Paroxetine When Used for the Treatment of Premenstrual Dysphoria
Brief Title: A Placebo-Controlled Study to Investigate the Onset of Action of Paroxetine in Premenstrual Dysphoria
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Novo Nordisk A/S (Industry); GlaxoSmithKline (Industry); Göteborg University (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: L&E-5
Record Dates: First submitted 2007-08-13; First posted 2007-08-14 (Estimated); Last update posted 2007-12-07 (Estimated); Status verified 2007-08

CONDITIONS: Premenstrual Dysphoric Disorder; Premenstrual Syndrome
Keywords: paroxetine; onset of action; serotonin reuptake inhibitors
MeSH Terms: conditions — Premenstrual Dysphoric Disorder; Premenstrual Syndrome | interventions — Paroxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Paroxetine 20mg during the luteal phase of the menstrual cycle
  Interventions: Drug: paroxetine
- 2 (Placebo Comparator): Placebo during the luteal phase of the menstrual cycle
  Interventions: Drug: paroxetine

INTERVENTIONS:
Drug: paroxetine — Capsules containing either placebo or paroxetine 20 mg. The treatment start after ovulation and when the subject has experienced premenstrual irritability for 2 days. The dosage is one capsule daily at 8 AM

SUMMARY:
The objective of this study is to explore the onset of action when serotonin reuptake inhibitors are used to treat premenstrual dysphoric disorder

DETAILED DESCRIPTION:
Whereas serotonin reuptake inhibitors (SRIs) usually require weeks of treatment to effectively counteract depressed mood or anxiety, several studies suggest that they may reduce the symptoms irritability and anger more rapidly. In line with this, SRIs have been shown to reduce certain symptoms, including irritability, in women with premenstrual dysphoric disorder (PMDD) when the drug only is administered from ovulation to menstruation only, which indicates an onset of action of 10 days or less. How fast this effect appears in terms of hours or days is, however, not known. The objective of this study was to explore this issue.

ELIGIBILITY:
Inclusion Criteria:

* The patient should have participated in an ongoing placebo-controlled trial regarding the effect of paroxetine in PMD; to be included in that trial, she must have fulfilled the diagnostic criteria A-C of PMDD in DSM-IV and certain other inclusion and exclusion criteria which are listed in appendix 1.
* The patient should a) have been given paroxetine during the previous trial, b) have reported that she has been "much improved" or "very much improved" by this treatment, c) have displayed a marked reduction in VAS-rated irritability during treatment, and d) have reported that she has found the side-effects tolerable.
* The patient should display at least a 50% increase in VAS-rated irritability during the luteal phase (mean of last five days prior to menses) as compared the follicular phase (days 6-10) during one cycle of pretreatment symptom rating (without medication).
* The patient should have given written informed consent to participate in the study.

Exclusion Criteria:

* Any concomitant psychiatric disorder for which SRIs are known to be effective.
* Any other concomitant psychiatric disorder that, in the investigator's opinion, would render the patient unsuitable for the study.
* Any somatic disorder that, in the investigator's opinion, would render the patient unsuitable for the study.
* Any ongoing medication which, in the opinion of the investigator, would render the patient unsuitable for the study. Examples of medications that preclude participation in the study are: 1) any psychotropic drug, with the exception of the occasional use of hypnotics, 2) any hormonal preparation, with the exception of thyroid hormone, 3) anti-coagulants, and 4) 5HT1D agonists. Occasional use of analgesic compounds does not preclude participation.
* Patient characteristics which, in the opinion of the investigator, are likely to reduce compliance with the protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2000-10; Study Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
The number of patients reaching sustained remission (irritability) for each time point

SECONDARY OUTCOMES:
Self rated irritability at each time point

CONTACTS AND LOCATIONS:
Overall Officials: Mikael SG Landen, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- The Psychiatric clinic, Sahlgrenska University Hospital, Gothenburg, Sweden